CLINICAL TRIAL: NCT00606866
Title: Dynamic-Contrast Enhanced MRI Pharmacodynamic Study of BAY 43-9006 in Metastatic Renal Cell Carcinoma
Brief Title: MRI Study of BAY 43-9006 in Metastatic Renal Cell Carcinoma
Acronym: MRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12977A
Record Dates: First submitted 2008-01-31; First posted 2008-02-05 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: renal, metastatic, carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Carcinoma | interventions — Sorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Placebo Comparator): placebo pill
  Interventions: Drug: placebo
- II (Active Comparator): Sorafenib, 200 mg bid
  Interventions: Drug: Sorafenib
- III (Active Comparator): Sorafenib, 400 mg bid
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: placebo — Placebo for four weeks
  Arms: I
Drug: Sorafenib — Sorafenib 200 mg twice daily
  Arms: II
Drug: Sorafenib — Sorafenib, 400 mg twice daily
  Arms: III

SUMMARY:
The purpose of this study is to determine maximum tumor shrinkage, time to progression, survival, drug concentration, and degree of skin toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic clear cell renal cell cancer;
* At least one lesion that can be accurately measured in at least one dimension;
* Patients must not have been treated with prior anti-timor kinase inhibitors or VEGF pathway inhibitors;
* Age 18 and older;
* ECOG performance status 0-2;
* Blood pressure higher than 140/90 on 2 separate occasions not more than 6 weeks prior to enrollment and not less than 24 hours apart;
* Normal organ function: total bilirubin less than upper limit of normal, AST less than 2.5 X upper limit of normal, creatinine less than 2.8 mg/dl;
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation;
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Chemotherapy or radiotherapy within 4 weeks prior to entering the study;
* Any other investigational agents;
* Known brain metastases;
* Uncontrolled intercurrent illness including ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-07; Primary Completion 2007-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To determine whether a new experimental MRI technique called "Dynamic Contrast Enhanced MRI" (DCE-MRI) can determine the best dose of sorafenib | 8 weeks

SECONDARY OUTCOMES:
To predict which patients are most likely to experience tumor shrinkage. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States